CLINICAL TRIAL: NCT06502340
Title: ASSESSMENT OF PERIOPERATIVE MYOCARDIAL DAMAGE IN ROBOT-ASSISTED LAPAROSCOPIC RADICAL PROSTATECTOMIES
Brief Title: PERIOPERATIVE MYOCARDIAL DAMAGE IN ROBOT-ASSISTED SURGERY
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, assoc. prof, Ankara City Hospital Bilkent
Other Study IDs: E2-23-5211
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Myocard Injury After Non Cardiac Surgery; Robotic Assisted Laparoscopic Radical Prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — high-sensitive Troponin I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: All patients who will undergo elective robotic-assisted laparoscopic radical prostatectomy
  Interventions: Diagnostic Test: high sensitive troponin I

INTERVENTIONS:
Diagnostic Test: high sensitive troponin I — high-sensitive Troponin I levels

SUMMARY:
Our study aimed to identify myocardial damage during or after robotic-assisted radical prostatectomy by measuring high-sensitive Troponin I levels, which are the most sensitive and effective according to the AHA/ACC guideline. The study's secondary objective was to establish which parameters were associated with myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective robotic surgery
* Patients with I, II, and III according to ASA classification
* Those with body mass index (BMI) below 35kg/m2
* Patients whose consent was obtained before the procedure

Exclusion Criteria:

* Patients who were converted to open surgery for any reason
* patients who did not agree to participate in the research

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing elective robotic-assisted laparoscopic radical prostatectomy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
high-sensitive Troponin I levels | preoperative
high-sensitive Troponin I levels | postoperative 24th hour
high-sensitive Troponin I levels | postoperative 48th hour

IPD SHARING:
Plan to Share IPD: Undecided